CLINICAL TRIAL: NCT06916754
Title: Comparing the Efficacy of Combined Behavioral Intervention and Ericksonian Hypnotherapy in the Treatment of Alcohol Addiction: A Randomized Controlled Trial
Brief Title: Comparing Combined Behavioral Intervention and Ericksonian Hypnotherapy for Alcohol Addiction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beykoz University (Other)
Collaborators: Istanbul Nisantasi University (Other); Uskudar University (Other)
Responsible Party: Principal Investigator, Eda Yilmazer, Principal Investigator, Beykoz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEYKOZ-EH-CBI-2025
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Alcohol-Related Disorders; Alcoholism; Substance-related Disorders
Keywords: Ericksonian Hypnosis; Hypnotherapy; Cognitive Behavioral Therapy; Motivational Interviewing; Relapse Prevention; Craving; Substance Craving; Psychotherapy
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Three-arm, parallel-group randomized controlled trial with equal allocation to Combined Behavioral Intervention (CBI), Ericksonian Hypnotherapy (EH), or control (standard care information). Each participant receives only one type of intervention throughout the 12-week treatment period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors who collect follow-up and post-treatment data will be blinded to participants' group assignment. Participants and therapists are not blinded due to the nature of behavioral interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Behavioral Intervention (CBI) (Experimental): Participants in this arm will receive a manualized Combined Behavioral Intervention consisting of 12 weekly sessions, each approximately 60 minutes. The intervention includes elements of Motivational Interviewing, Cognitive Behavioral Therapy, and relapse prevention strategies. Sessions are delivered either individually by licensed therapists trained in behavioral therapy.
  Interventions: Behavioral: Combined Behavioral Intervention
- Ericksonian Hypnotherapy (EH) (Experimental): Participants in this arm will receive Ericksonian Hypnotherapy in 12 weekly individual sessions, each approximately 45-60 minutes. The intervention uses personalized trance induction, metaphorical storytelling, ego-strengthening, and post-hypnotic suggestions.
  Interventions: Behavioral: Ericksonian Hypnotherapy
- Control (Standard Care Information) (No Intervention): Participants in this group will not receive structured psychotherapy but will be provided with psychoeducational brochures and referral resources related to alcohol addiction treatment. They will complete the same assessment schedule as the other groups.

INTERVENTIONS:
Behavioral: Combined Behavioral Intervention — The intervention includes 12 weekly sessions integrating Motivational Interviewing, Cognitive Behavioral Therapy, and relapse prevention strategies. Techniques include enhancing motivation to change, identifying cognitive distortions, managing high-risk situations, and developing alternative coping strategies.
  Arms: Combined Behavioral Intervention (CBI)
Behavioral: Ericksonian Hypnotherapy — This therapy includes 12 weekly sessions involving individualized trance induction, indirect suggestion, therapeutic metaphor, and ego-strengthening techniques. The sessions follow Ericksonian principles and are delivered by certified hypnotherapists.
  Arms: Ericksonian Hypnotherapy (EH)

SUMMARY:
This clinical study is being conducted to compare the effectiveness of two psychological treatments for alcohol addiction: Combined Behavioral Intervention (CBI) and Ericksonian Hypnotherapy (EH). The purpose of the study is to determine whether Ericksonian Hypnotherapy, a more personalized and indirect therapeutic method, is equal to or more effective than the gold-standard approach, Combined Behavioral Intervention, in helping individuals reduce their alcohol consumption and improve psychological well-being.

Alcohol addiction is a serious condition that affects mental, emotional, and physical health. Many treatment options exist, but not all individuals respond in the same way. This study aims to evaluate two different types of therapy in a structured way, to better understand which works best, for whom, and under what circumstances.

The study will include 90 adult participants diagnosed with Alcohol Use Disorder (AUD). Participants will be randomly assigned to one of three groups: (1) a group receiving weekly sessions of Combined Behavioral Intervention, (2) a group receiving weekly sessions of Ericksonian Hypnotherapy, or (3) a control group receiving general educational materials about alcohol addiction. Treatment will last for 12 weeks, and all participants will be followed up three months after the last session to assess long-term effects.

Throughout the study, researchers will measure changes in alcohol consumption, alcohol craving, mental health symptoms (such as depression and anxiety), quality of life, and motivation to change. The findings of this study may help improve the way alcohol addiction is treated by offering evidence on alternative approaches such as hypnotherapy.

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) is a persistent and relapsing condition with profound personal, familial, and societal consequences. Although several psychosocial interventions have demonstrated efficacy, there remains an unmet need for alternative, accessible, and effective therapeutic approaches that can be tailored to individual needs and cognitive styles. Combined Behavioral Intervention (CBI), which integrates Motivational Interviewing (MI), Cognitive Behavioral Therapy (CBT), and relapse prevention strategies, is regarded as a gold-standard modality for the treatment of alcohol addiction. Ericksonian Hypnotherapy (EH), in contrast, represents a less traditional but increasingly recognized intervention that uses indirect suggestion, personalized metaphor, and trance-based language to target the unconscious processes that often underlie maladaptive behaviors such as substance use.

This randomized controlled trial (RCT) aims to directly compare the clinical efficacy of CBI and EH in reducing alcohol use and related psychological symptoms among adults diagnosed with AUD. The trial also seeks to assess differential impacts on craving typologies, cognitive beliefs related to addiction, mental health symptoms, quality of life, and motivation to change. While CBI is grounded in conscious, structured therapeutic engagement and skill acquisition, EH offers a fluid and individualized therapeutic experience that may bypass conscious resistance, making it especially relevant for individuals who struggle with conventional, didactic approaches.

A total of 90 adult participants will be enrolled, all of whom will meet DSM-5 diagnostic criteria for Alcohol Use Disorder (mild to severe), confirmed by a qualified psychiatrist. Participants will be recruited through private psychiatric clinics and general psychiatry outpatient services in Istanbul, Turkey, leveraging a network of collaborating clinicians who will refer eligible individuals. After informed consent and baseline screening, participants will be randomly assigned in equal numbers (1:1:1) to one of three study arms: (1) Combined Behavioral Intervention (CBI), (2) Ericksonian Hypnotherapy (EH), or (3) control group receiving general educational materials and referral guidance without structured psychotherapy.

Participants in the CBI group will attend 12 weekly individual or small group sessions (depending on scheduling and logistics), each lasting approximately 60 minutes. These sessions will systematically cover motivation enhancement, cognitive restructuring, coping with triggers, and relapse prevention strategies. The EH group will also receive 12 weekly sessions lasting approximately 45-60 minutes each. These sessions will employ individualized hypnotic induction techniques, ego-strengthening interventions, post-hypnotic suggestions, and metaphoric storytelling designed to promote subconscious readiness for change. Audio recordings will be provided to support daily self-hypnosis practice at home, though this is not mandatory. The control group will receive psychoeducational materials related to alcohol addiction, as well as referral contact information for local support services, but will not engage in any structured therapeutic process.

The study will involve repeated measurement of both behavioral and psychological variables across four timepoints: baseline (T0), midpoint of treatment at Week 6 (T1), post-treatment at Week 12 (T2), and follow-up at Month 10 (T3). The primary outcome is alcohol consumption, measured by the Timeline Follow-Back (TLFB) method-a validated, retrospective self-report tool assessing daily drinking over the past 30 days.

Secondary outcomes include both cognitive and phenomenological dimensions of craving, measured using the Craving Beliefs Questionnaire (CBQ) and the Craving Typology Questionnaire (CTQ), respectively. These instruments offer a dual lens into the subjective experience of craving: CBQ focuses on belief systems that maintain substance use (e.g., perceived uncontrollability), while CTQ distinguishes between obsessive, relief-oriented, and reward-based craving patterns. Depression and anxiety symptoms will be assessed using either the Beck Depression Inventory-II (BDI-II) or Patient Health Questionnaire-9 (PHQ-9) and the Beck Anxiety Inventory (BAI) or Generalized Anxiety Disorder-7 (GAD-7), depending on participant suitability and assessment availability. Broader quality-of-life impacts will be measured using the WHO Quality of Life-BREF (WHOQOL-BREF) or alternatively the Short Form-12 (SF-12). Readiness to change will be assessed with the Turkish version of the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES).

Adherence to treatment (session attendance) and participant satisfaction with therapy will also be recorded, alongside reasons for withdrawal if applicable. Outcome data will be collected and coded by trained, blinded assessors who will have no role in therapy delivery or treatment group assignment.

Statistical analysis will follow an intention-to-treat (ITT) principle. The primary outcome-change in alcohol consumption-will be analyzed using linear mixed-effects modeling or repeated measures ANOVA with fixed effects for group, time, and group-by-time interactions. Secondary analyses will explore group differences in craving, mental health symptoms, and readiness to change using similar longitudinal methods. Multiple imputation or last observation carried forward (LOCF) strategies will be employed to address missing data. Subgroup analyses based on baseline severity and comorbidity may be conducted if sample size permits.

The central hypothesis of the study is that Ericksonian Hypnotherapy will be non-inferior or superior to Combined Behavioral Intervention in reducing alcohol use and related craving. It is further hypothesized that while CBI will lead to stronger improvements in belief-driven cognitive mechanisms, EH may be more effective in addressing the emotional and phenomenological dimensions of craving. Both active treatments are expected to yield superior outcomes compared to the control group.

By testing a structured comparison between a widely used evidence-based model (CBI) and a less conventional yet promising method (EH), this study has the potential to inform clinical decision-making, diversify treatment options, and contribute new insights into how psychological and hypnotic methods can be integrated into substance use treatment. The use of both cognitive and experiential craving assessments, together with validated instruments and a robust design, supports the methodological rigor of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Meets DSM-5 diagnostic criteria for Alcohol Use Disorder (mild to severe)
* Medically and psychiatrically stable as determined by a clinician
* Willing and able to participate in weekly sessions over a 12-week period
* Provides informed consent

Exclusion Criteria:

* Current diagnosis of a severe psychiatric disorder (e.g., psychotic disorder, bipolar I disorder)
* Significant cognitive impairment that would interfere with treatment participation
* Participation in another structured addiction treatment during the study period
* Current use of psychotropic medications that may influence outcome measures (as assessed by the clinical team)
* Unstable medical condition requiring immediate intervention
* Pregnancy or planning to become pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Consumption (TLFB) | Baseline to Week 6, Week 12, and Month 10 (3-Month Follow-Up)
  Self-reported alcohol consumption measured using the Timeline Follow-Back (TLFB) method. TLFB assesses the number of standard drinks consumed each day over the past 30 days. Higher scores indicate greater alcohol use. A reduction in total drinks consumed per month represents clinical improvement.

SECONDARY OUTCOMES:
Change in Craving Beliefs (CBQ) | Baseline to Week 6, Week 12, and Week 24
  Craving Beliefs Questionnaire (CBQ) measures dysfunctional beliefs about alcohol craving. Scores range from 20 to 140, with higher scores indicating more maladaptive craving-related beliefs. A reduction in CBQ scores indicates improvement.
Change in Craving Typologies (CTQ) | Baseline to Week 6, Week 12, and Week 24
  Craving Typology Questionnaire (CTQ) measures three dimensions of craving: obsessive, relief, and reward craving. Each subscale ranges from 0 to 36, with higher scores indicating greater craving intensity. Reductions in subscale scores reflect improvement.
Change in Depression Symptoms (BDI-II) | Baseline to Week 6, Week 12, and Week 24
  Depressive symptoms assessed using either the Beck Depression Inventory-II (range: 0-63). Higher scores indicate more severe depression. A decrease in total score reflects symptom improvement.
Change in Anxiety Symptoms (BAI) | Baseline to Week 6, Week 12, and Week 24
  Anxiety symptoms measured with the Beck Anxiety Inventory (range: 0-63). Higher scores reflect greater anxiety severity. A reduction in total score indicates clinical improvement.
Change in Quality of Life (WHOQOL-BREF) | Baseline to Week 6, Week 12, and Week 24
  Measured using the WHOQOL-BREF (domain scores range from 4 to 20, with higher scores indicating better quality of life). Increases in scores represent improved well-being.
Change in Readiness to Change (SOCRATES) | Baseline to Week 6, Week 12, and Week 24
  SOCRATES measures motivation to change alcohol use behavior across three dimensions: Recognition, Ambivalence, and Taking Steps. Subscales range from 7 to 35. Higher scores represent greater readiness to change. Improvements reflect increased motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Gökben Hızlı Sayar, Prof, Study Chair — Üsküdar University; Selami Varol Ülker, Phd, Study Director — Üsküdar University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University
Locations (1):
- Beykoz University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in published articles will be shared. This includes data on alcohol use, craving (CBQ and CTQ), depression, anxiety, quality of life, motivation to change, and session attendance. Data will be made available to qualified researchers affiliated with academic or nonprofit institutions upon request and approval. Data will be shared through secure institutional repositories.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available upon request starting immediately after the publication of the main study findings in a peer-reviewed journal. Data will remain accessible for 36 months after the date of publication.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or non-profit institutions who provide a methodologically sound proposal approved by the study team. Requesters must sign a data use agreement. Access will include de-identified individual participant data and supporting documents. Requests can be submitted via email to the principal investigator following publication.